CLINICAL TRIAL: NCT07034196
Title: Comparative Effectiveness of Primary Care Providers Trained in Rheumatoid Arthritis Management Versus Rheumatologist Care: A Randomized Controlled Trial
Acronym: TRAIN
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: St. Lawrence Health System (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro00080017; TRMAA (Other: NYS Vital Access Provider MCD)
Record Dates: First submitted 2025-06-13; First posted 2025-06-24 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-06

CONDITIONS: Rheumatoid Arthritis (RA
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Arm- Rheumatology Clinician (No Intervention): Continue with usual RA care in their rheumatologist's office
- Intervention Arm- Primary Care Clinician (Active Comparator): RA patients will be randomized to receive their RA care via their established PCP who completed a structured training course in RA and who has monthly case review/consultation sessions with the rheumatology team in this study
  Interventions: Other: Primary Care Treatment in lieu of Rheumatologist

INTERVENTIONS:
Other: Primary Care Treatment in lieu of Rheumatologist — RA patients will be randomized to receive their RA care via their established PCP who completed a structured training course in RA and who has monthly case review/consultation sessions with the rheumatology team in this study
  Arms: Intervention Arm- Primary Care Clinician

SUMMARY:
Rheumatoid arthritis (RA) is a complex autoimmune disease where the immune system attacks healthy joint tissue; causing pain, swelling, and stiffness of the joints. This disease effects lots of people in the US and can lead to major joint damage if not properly treated. In rural areas like northern NY, these are underserved areas for RA patients, thus many patients struggle to get the appropriate care. This model is testing whether primary care providers (PCP) can safely and effectively provide stable RA patients with the proper treatment rather than send them to a specialist. PCPs were trained through classes, case reviews, and a final exam. Patients will be randomly assigned to either see a trained PCP or their normal rheumatologist at the rheumatology clinic. This study will examine how patients are doing over a year using medical exams and patient feedback. If this model proves to be successful, it will make RA treatment easier and more affordable for patients.

DETAILED DESCRIPTION:
Rheumatoid arthritis (RA) is a chronic autoimmune disorder characterized by joint inflammation, stiffness, and pain. If left untreated, RA can lead to irreversible joint damage and functional impairment. This disease has significant impact on the healthcare system of the United States because it requires specialized care, while also affection about 1.5 million individuals [Pfizer, 2025]. Within the United States, access to specialized care is not widespread, with large disparities between urban and rural areas. Rural areas have about 1/8th the specialists per 100,000 people when compared to urban areas [NRHA]. Access to timely and effective care is vital to maintain the quality of life of RA patients. St. Lawrence Health (SLH) is a rural health system in St. Lawrence County in northern New York. SLH not only serves its own county, but the four surrounding counties. Eyal Kedar, MD, is the sole rheumatologist of this expansive region, and manages a large RA patient load. If there were more access to RA management in our area, our rheumatology clinic would be more available for patients who need to see a rheumatologist for something other than RA.

This trial will evaluate if trained primary care providers (PCPs) can give care that is meets the standards set by our rheumatology clinic. Nine PCPs in our area were selected and subjected to a structured training course involving regularly scheduled lectures, discussions, case studies and a final exam to test the knowledge obtained through these training sessions. The trial will consist of two arms, the intervention arm (Arm 1) and the active comparator (control) arm (Arm 2). In Arm 1, patients will be seeing their established PCP who has completed the RA training for their RA management. In Arm 2, patients will be meeting with our rheumatology clinic with either a rheumatologist or a rheumatology APP. Patients will be randomly assigned to one of these arms in a 1:1 ratio. Maximum enrollment of this trial is one hundred subjects, and PCPs will see a minimum of two subjects and a maximum of twenty. Over the course of the study, there will be monthly case review sessions with the rheumatology team, and ad hoc consultations outside of the monthly meeting as needed. The study will collect data at screening/baseline, 6 weeks, 12 weeks, 26 weeks, 40 weeks, and 52 weeks utilizing standard assessments of RA activity (MD_HAQ, Evaluator Global assessment, Tender and Swollen Joint Count, DAS28 Calculation, CDAI Calculation, and SDAI Calculation, Glucocorticoid Exposure), patient-reported outcomes and medical records review.

If the study shows PCP's that are properly trained can effectively manage stable RA patients, this could vastly improve chronic disease management in underserved areas like the northern country of New York State. This model would allow healthcare systems to better utilize workforce capacity, reduce burden on subspeciality care, and possibly lower cost associated with receiving treatment. Furthermore, the success could be applicable to other complex chronic diseases like lupus, chronic kidney disease, etc. This would serve as the blueprint for sustainable and scalable care that would meet the needs of patients in the rural areas without relying on telemedicine or other forms of treatment.

For patients, especially those living in remote areas, the benefits of this study would be significant. If the model was to be successful, it would eliminate the need for long-distance driving to specialists, make it more affordable and easier to receive care in a timely manner. Patients would have the benefit of receiving care from their trusted PCP who are trained by the rheumatology department. This would allow for better disease control, a better quality of life, and possibly great satisfaction with the treatment given. Furthermore, this model will enhance overall health care in the northern country as by expanding the pool of providers that are able to manage complex diseases.

This trial is a pioneering effort to more efficiently deal with chronic disease care in rural areas. By training PCPS to take a lead in RA management, this study may offer a possible solution to the subspecialty shortages that effect millions of rural residents. Thus, if this model proves to be successful, this will not only better the lives of RA patients in the rural areas but will pave the way for more efficient healthcare delivery methods across the world.

ELIGIBILITY:
Inclusion Criteria:

* Fulfillment of the 2010 ACR/EULAR classification criteria for rheumatoid arthritis Using these criteria, a classification as "definite RA" is based upon the presence of synovitis in at least one joint, the absence of an alternative diagnosis that better explains the synovitis, and the achievement of a total score of at least 6 (of a possible 10) from the individual scores in four domains.

The highest score achieved in a given domain is used for this calculation. These domains and their values are:

* Number and site of involved joints:

  * 2 to 10 large joints (from among shoulders, elbows, hips, knees, and ankles) = 1 point
  * 1 to 3 small joints (from among the MCP joints, PIP joints, second through fifth MTP joints, thumb IP joints, and wrists) = 2 points
  * 4 to 10 small joints = 3 points
  * Greater than 10 joints (including at least 1 small joint) = 5 points
* Serological abnormality (RF or ACPA)

  * Low positive (above the upper limit of normal) = 2 points
  * High positive (greater than three times the upper limit of normal) = 3 points
* Elevated acute phase response (ESR or CRP) above the upper limit of normal = 1 point
* Symptom duration at least six weeks = 1 point

  * Stable disease activity, defined as a RAPID-3 score of no higher than 4 over the past three months or no RA-related medication changes for at least six months prior to the informed consent date.
  * Primary residence in the North Country region of New York (Jefferson, Lewis, St. Lawrence, Clinton, Essex, Franklin, and Hamilton counties).
  * Established with the participating rheumatology clinic and a participating PCP (Note: For patients who are established in PCP clinics outside of the health system conducting this study, patients may see a participating PCP within their established clinic). To be considered an established patient, the participant should have had a visit within the year prior to the screening visit.
  * Willingness to participate in the study and provide informed consent.
  * Females of childbearing potential must agree to use highly effective birth control throughout duration of the study.

Exclusion Criteria:

* Changes in RA treatment within the six months prior to screening.
* History of interstitial lung disease or any manifestation of rheumatoid vasculitis including cutaneous rheumatoid vasculitis, vasculitic neuropathy, RA-associated episcleritis, scleritis or keratitis)
* Cognitive impairment or inability to complete study assessments.
* Pregnancy, breastfeeding, or plans to become pregnant during the study period.
* Inability to adhere to the study protocol or follow-up requirements.
* Any comorbid condition that, in the opinion of the investigator, would make the subject unsuitable for participation in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-06-26 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in Disease Activity Score (DAS-28) | 6 and 12 month intervals relative to baseline
  The primary efficacy endpoint is the change in Disease Activity Score (DAS-28) response at 6 and 12 month intervals relative to baseline. It will be evaluated for non-inferiority of the treatment effect. The treatment difference between the Primary Care group and the Rheumatology group may be presented with point estimate and 95% CI.

CONTACTS AND LOCATIONS:
Overall Officials: Eyal Kedar, MD, Principal Investigator — St. Lawrence Health
Locations (1):
- St. Lawrence Health, Potsdam, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Battafarano DF, Ditmyer M, Bolster MB, Fitzgerald JD, Deal C, Bass AR, Molina R, Erickson AR, Hausmann JS, Klein-Gitelman M, Imundo LF, Smith BJ, Jones K, Greene K, Monrad SU. 2015 American College of Rheumatology Workforce Study: Supply and Demand Projections of Adult Rheumatology Workforce, 2015-2030. Arthritis Care Res (Hoboken). 2018 Apr;70(4):617-626. doi: 10.1002/acr.23518. PMID 29400009